CLINICAL TRIAL: NCT06036524
Title: Development and Identification of Magnetic Resonance, Electrophysiological, and Fiber-optic Imaging Biomarkers of Myofascial Pain
Brief Title: Multi-modal Imaging of Myofascial Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202201039; R61AT012283 (NIH)
Record Dates: First submitted 2023-08-08; First posted 2023-09-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Myofascial Pain
Keywords: Magnetic Resonance Imaging; Surface Electromyography; Fiber-optic Imaging and Sensing

STUDY DESIGN:
Intervention Model Description: This is a two-phase, NIH-supported study. The first R61 phase (currently awarded) is an observational study with one control group and one patient group. The second R33 phase is a randomized clinical trial, which will be awarded by the end of the R61 phase. The study design provided here is for R61 only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-modal imaging of myofascial pain (Experimental): Participants with and without myofascial-related pain disease will receive multi-modal, multi-parametric, multi-scale imaging, including magnetic resonance imaging, surface electromyography, and fiber-optic imaging and sensing.
  Interventions: Diagnostic Test: Multi-modal, multi-parametric, multiscale imaging of the myofascial unit

INTERVENTIONS:
Diagnostic Test: Multi-modal, multi-parametric, multiscale imaging of the myofascial unit — Study Participants will undergo four study procedures at one visit, including magnetic resonance imaging (MRI), surface electromyography (sEMG), fiber-optic imaging and sensing, and questionnaires.

SUMMARY:
The goal of this study is to develop new imaging biomarkers for quantitative assessments of myofascial pain.

DETAILED DESCRIPTION:
This study aims to develop a multi-modal, multi-parametric, multi-scale imaging of the human myofascial unit by combining magnetic resonance imaging (MRI), surface electromyography (sEMG), and fiber-optic imaging and sensing.

Participants (half with active neck/shoulder/back pain, and half healthy controls) will be recruited from pain management clinics and Volunteer for Health, or will be referred by Dr. Xioabin Yi. They will undergo all three imaging techniques and complete a number of patient questionnaires over the course of a single study visit. The study team will then identify candidate biomarkers capable of differentiating between healthy (no myofascial pain) and those with active pain to target in a future clinical trial.

ELIGIBILITY:
Healthy Volunteer Inclusion Criteria:

1. Absence of a history of chronic pain in the targeted anatomical location (i.e., neck and shoulder) that had limited activities of daily living or work
2. A numerical current pain index of lower than 0.5 according to initial assessment with visual analog scale
3. Able to understand the goal of the project and give informed consent.

Healthy Volunteer Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Contraindication to MRI
3. Previous severe/acute neck or shoulder injury
4. Previous neck or shoulder surgery
5. Neck or shoulder deformities
6. Inability to provide consent.

Myofascial Pain Patient Inclusion Criteria:

1. Between the ages of 18 and 80 years old
2. Neck and/or shoulder pain, unilateral or bilateral
3. Duration of symptoms for longer than 4 weeks
4. Pain scale at the active state higher than 4 according to initial assessment with visual analog scale
5. Presence of active trigger point(s) according to palpation and/or presence of taut band

Myofascial Pain Patient Exclusion Criteria:

1. Recent history of trauma to the neck (e.g., whiplash)
2. Acute cervical radiculopathy
3. Acute cervical spine pain component or acute cervical spinal pathology Presence of neuromuscular pathologies or inflammatory muscle diseases (e.g., dermatomyositis)
4. Systemic disease with diffuse body pain (e.g., system lupus erythematosus and and thyroid disease)
5. Peripheral neuropathy
6. Cancer-related pain
7. Pregnancy, coagulopathy, fever, general/local infection at the pain site, substance abuse, peripheral neuropathy, or any other diseases that may account for signs and symptoms mimicking myofascial pain
8. Contraindication to MRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Statistical Plan | For each individual, multi-modal imaging will be performed on the same day. Magnetic Resonance Imaging (MRI) will take about 1 hour. Fiber-optic measurements will take a few minutes. Surface electromyography (sEMG) recording will take <20 minutes.
  The statistical analysis will assess the capability of imaging-based quantitative biomarkers to distinguish the pathological and physiological differences between participant groups (i.e., myofascial pain patients vs. healthy volunteers). The imaging biomarkers will be measured for each participant, including tissue stiffness, hydration, inflammation, blood oxygenation and flow, electrical activity, etc. The biomarkers will be measured and compared in the univariate fashion, which means we assess the differentiation performance for each biomarker independently. For each biomarker, we will compare the difference between the participant groups, using the Student's t-test or Wilcoxon rank-sum test. The statistical power will be estimated based on the effect size (Cohen's d) of difference between the participant groups. With an expected effect size of >0.9, the proposed sample size can achieve a statistical power greater than 0.8.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No